CLINICAL TRIAL: NCT02874209
Title: Noninvasive Assessment of Neuronal Damage by MRI Sodium ( 23Na ) in Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015-15; 2015-A00328-41 (Other: Ansm)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient with amyotrophic lateral sclerosis (Experimental): ALS patients with, spinal and bulbar form, certain or probable diagnosis according to the revised El Escorial criteria will go through the MRI sodium
  Interventions: Other: sodium MRI
- Healthy volunteer (Placebo Comparator): Healthy Volonteer apparied for sexe and age with selected ALS patients will go through the MRI sodium
  Interventions: Other: sodium MRI

INTERVENTIONS:
Other: sodium MRI

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease affecting the central and peripheral motor neurons, characterized by the rapidity of its evolution (median survival of 3 years). The pathophysiology of the disease is still poorly understood. Neuronal death results from several cellular mechanisms entangled, including mitochondrial dysfunction. The absence of diagnostic marker causes a significant delay in diagnosis, on average a year. On the other hand, the wish biomarker is important for therapeutic trials. Recently, MRI sodium (23Na) demonstrated its importance to detect noninvasively sodium accumulations associated with neuronal suffering. This neuronal pain can be caused by mitochondrial dysfunction causing the accumulation in the sodium and calcium cell causing neuronal death. These studies were conducted in multiple sclerosis, Alzheimer's disease, Huntington's disease, stroke and brain tumors. They demonstrated that sodium MRI could be an effective and sensitive biomarker for detecting and quantifying neuronal degeneration. The goal of this study is to assess neuronal damage noninvasively by MRI sodium in amyotrophic lateral sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic lateral sclerosis patient according to the El Escorial criteria revised Brooks et al. 2000 bulbar or spinal beginning

Exclusion Criteria:

* patient or healthy volonteer presenting MRI contre indications to this exam.
* patient or healthy volonteer presenting severe high blood pressure undergoing medication to treat it or not.
* patient or healthy volonteer having chronic psychiatric illness, dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Central conduction time of the potential muscle through transcranial magnetic stimulation | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Urielles DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille; Aude GRAPPERON, Md, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Masreille, France

IPD SHARING:
Plan to Share IPD: No